CLINICAL TRIAL: NCT00914797
Title: Blood and Urinary Concentrations of Terbutaline in Asthmatics and Elite Athletes With Asthma: Comparison Between Inhalation vs. Oral Administration.
Brief Title: Terbutaline Concentrations in Blood and Urine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other)
Responsible Party: Jimmi Elers, Respiratory Research Unit, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: TER2009JE
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
Keywords: Asthma; Doping; Beta agonist; Terbutaline; Pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — Inhalation; Terbutaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- asthmatics (Active Comparator): 10 male asthmatic subjects
  Interventions: Drug: inhaled and oral terbutaline
- healthy (Active Comparator): 10 male healthy volunteers
  Interventions: Drug: inhaled and oral terbutaline
- elite athletes with asthma (Active Comparator): 10 elite athletes with asthma.
  Interventions: Drug: inhaled and oral terbutaline

INTERVENTIONS:
Drug: inhaled and oral terbutaline — Inhalation of 2 mg terbutaline as powder as a single dosage. Oral terbutaline 10 mg as a single dosage.
  Inhaled: Bricanyl Turbohaler 0.5 mg/dose, MA no. 41076.
  Oral: Tablet Bricanyl Retard 5 mg, MA no. 10954.
  Other Names: Bricanyl Turbohaler 0.5 mg/dose, MA no. 41076.; Tablet Bricanyl Retard 5 mg, MA no. 10954.

SUMMARY:
The purpose of this study is to assess the blood and urine concentrations of terbutaline and to evaluate the difference between inhaled and oral terbutaline in order to distinguish treatment with terbutaline from doping with terbutaline in a doping control.

DETAILED DESCRIPTION:
To investigate the serum and urine concentrations of terbutaline and evaluate the difference between inhaled terbutaline (2 mg) and oral terbutaline (10 mg) in order to distinguish doping with terbutaline from anti-asthmatic treatment with terbutaline.

To investigate the above mentioned in three groups: healthy men, male asthmatic subjects and male elite athletes with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma with positive reversibility or challenge test.
* Informed consent.
* Age between 18 - 45 years.
* Sex: male.
* Asthma classified as mild to moderate according to GINA guidelines.
* Used beta-2-agonist in minimum 12 months.

Exclusion Criteria:

* Smokers or ex-smokers with a smoking history of 10 pack years or more.
* Respiratory tract infections within the last 2 weeks prior to visit 1 and 2.
* Subjects with other chronic diseases than asthma and allergy.
* Allergy towards the study medicine.
* Use of beta-2-agonist 6 days prior to study day.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Terbutaline concentrations in serum and urine | baseline, 4, 8, and 12 hours after medicine administration

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Elers, MD, Principal Investigator — Bispebjerg Hospital, Respiratory Research Unit
Locations (1):
- Bispebjerg Hospital, Respiratory Research Unit, København NV, Denmark